CLINICAL TRIAL: NCT05434624
Title: The Effect of Bispectral Index Controlled Sedation on QT Distance and P Dispersion in ECG in Patients Having Bronchoscopy in the Intensive Care Unit
Brief Title: QT Distance and P Dispersion in ECG in Patients Having Bronchoscopy in the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Emine Ozsari, Assistant professor, Medical Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAIBU-MF-GH-EO-001
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Ventilator-Induced Lung Injury; Pulmonary Atelectasis
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Pulmonary Atelectasis | interventions — Midazolam; Propofol

STUDY DESIGN:
Intervention Model Description: For this study, it was planned to recruit 40 patients who would have FOB in the ICU of Abant İzzet Baysal University Anesthesia. All intubated patients over 18 years of age who do not meet the exclusion criteria will be included. Volume-controlled ventilation modes will be preferred during FOB. The pre-trade-inspired FiO2 will be increased to 100%. During the procedure, mean blood pressure, heart rate, oxygen saturation, respiratory rate, CVP, airway pressure, and BIS will be closely monitored. Enteral feeding will be discontinued at least 6 hours before the procedure. At the end of the procedure, the endotracheal tube position will be checked.
  FOB will be performed using mobile bronchoscopy (Storz FB; 5.0 mm outer diameter). All patients will be monitored with BIS (Bispectral Index A-2000, Aspect Medical Systems, Netherlands) to measure the depth of sedation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Experimental): Bronchoscopy group in which only midazolam will be used
  Interventions: Drug: Midazolam
- Group P (Experimental): Bronchoscopy group in which midazolam and propofol will be used
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Before the procedure, all patients were given i.v. 0:02 - 0:04 mg / kg midazolam (zolamide 15 mg / 3 mL, and medications, Turkey) will be administered.
  Other Names: Zolamid
  Arms: Group M
Drug: Propofol — Propofol 0.5 mg/kg bolus dose will be administered to Group II. Maintenance will be provided with 60 mcg/kg/min propofol infusion, and the propofol infusion dose will be increased by 10 mcg/kg/min by titration until the BIS value is 40-60 during the procedure.
  Other Names: Dormofol
  Arms: Group P

SUMMARY:
Fiberoptic bronchoscopy (FOB) is one of the most useful procedures for diagnosing and treating respiratory illnesses to figure out symptoms like hemoptysis, wheezing, or cough. Furthermore, FOB is a frequent method, in intensive care units, for both diagnoses of ventilator-associated pneumonia (VAP) and treatment of atelectasis with bedside sedation.) Propofol is often used in anesthesia for endoscopic treatments. Using propofol for deep anesthesia may be indicated to prevent the patient from feeling discomfort before FOB and to reduce the chance of complications.

Although major complications of FOB such as hypoxia and pneumothorax are known, there are limited studies showing its effects on cardiac hemodynamics. The cardiac effects of laryngoscope and intubation were investigated by using different anesthetic agents. In this study, we evaluated the effect of bronchoscopy with BIS-controlled sedation on ECG in ICU patients by monitoring the QT interval and P interval.

DETAILED DESCRIPTION:
For this study, it was planned to recruit 40 patients who would have FOB in the ICU of Abant İzzet Baysal University Anesthesia department. All intubated patients over 18 years of age who do not meet the exclusion criteria will be included. Before the procedure, all patients were given i.v. 0:02 - 0:04 mg / kg midazolam (zolamide 15 mg / 3 mL, and medications, Turkey) will be administered. Volume-controlled ventilation modes will be preferred during FOB. The pre-trade-inspired FiO2 will be increased to 100%. During the procedure, mean blood pressure, heart rate, oxygen saturation, respiratory rate, CVP, airway pressure, and BIS will be closely monitored. Enteral feeding will be discontinued at least 6 hours before the procedure. At the end of the procedure, the endotracheal tube position will be checked.

FOB will be performed using mobile bronchoscopy (Storz FB; 5.0 mm outer diameter). All patients will be monitored with BIS (Bispectral Index A-2000, Aspect Medical Systems, Netherlands) to measure the depth of sedation. Patients will be randomly divided into two groups by an anesthesiologist blinded to the study. Propofol will not be given to Group I after midazolam, while propofol 0.5 mg/kg bolus dose will be administered to Group II. Maintenance will be provided with 60 mcg/kg/min propofol infusion, and the propofol infusion dose will be increased by 10 mcg/kg/min by titration until the BIS value is 40-60 during the procedure. Patients under the age of 18, pregnancy, using sedative drugs in the last 24 hours, hypersensitivity to the drugs used in the study, severe cardiac disorder (EF: < 40), those who increase the QT interval (quinidine, lithium, procainamide, amiodarone, sotalol, phenothiazine, tricyclic Those who use antidepressants, disopyramide) or reducing (digitals) drugs, affecting QT such as hypomagnesemia- hypocalcemia - hypo or hyperthermia - hypo or hypercalcemia - hyperkalemia - hyper or hypothyroidism - myocarditis - mitral heart prolapse, etc. will be excluded from the study.

Patients will be randomly divided into 2 equal groups using the closed envelope method. Oral and written consent will be obtained from the first-degree relatives of all patients. All patients will be monitored with BIS to measure the depth of sedation. Age, weight - height, gender, medications used, comorbidities, hospitalization diagnosis, and duration of the procedure will be recorded for both groups. In addition, systolic blood pressure, diastolic blood pressure, mean blood pressure, heart rate, SpO2, BIS, respiratory rate, CVP, and airway pressure will be noted before and after the procedure of the first, fifth, tenth, and fifteenth minute. P wave dispersion, OTc, and OTd values will be calculated according to the max and min wavelengths as the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All intubated patients over 18 years of age

Exclusion Criteria:

* Patients under the age of 18
* Pregnancy
* Patients using sedative drugs in the last 24 hours
* Hypersensitivity to the drugs used in the study
* Severe cardiac disorder (EF: < 40)
* Patients using drugs that increase the QT interval (quinidine, lithium, procainamide, amiodarone, sotalol, phenothiazine, tricyclic antidepressants, disopyramide) or reduce the QT interval (digitals)
* Patients who have hypomagnesemia- hypocalcemia - hypo or hyperthermia - hypo or hypercalcemia - hyperkalemia - hyper or hypothyroidism - myocarditis - mitral heart prolapsus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
P wave dispersion (PWD) | Before the procedure
  PWD in all leads will be measured manually with the X10 magnifying glass. The beginning of the P wave is the point where the isoelectric line and the P wave intersect. The endpoint was taken as the intersection of the isoelectric line and the end point of the P wave.ECG recordings of at least 6 QRS for each lead
  1 mV at a rate of 20 mm/s, including the complex 3 channels in amplitude and standard 12 leads will be done simultaneously.
P wave dispersion (PWD) | After the procedure of the first minute
  PWD in all leads will be measured manually with the X10 magnifying glass. The beginning of the P wave is the point where the isoelectric line and the P wave intersect. The endpoint was taken as the intersection of the isoelectric line and the end point of the P wave.ECG recordings of at least 6 QRS for each lead 1 mV at a rate of 20 mm/s, including the complex 3 channels in amplitude and standard 12 leads will be done simultaneously.
P wave dispersion (PWD) | After the procedure of the fifth minute
  PWD in all leads will be measured manually with the X10 magnifying glass. The beginning of the P wave is the point where the isoelectric line and the P wave intersect. The endpoint was taken as the intersection of the isoelectric line and the end point of the P wave.ECG recordings of at least 6 QRS for each lead 1 mV at a rate of 20 mm/s, including the complex 3 channels in amplitude and standard 12 leads will be done simultaneously.
P wave dispersion (PWD) | After the procedure of the tenth minute
  PWD in all leads will be measured manually with the X10 magnifying glass. The beginning of the P wave is the point where the isoelectric line and the P wave intersect. The endpoint was taken as the intersection of the isoelectric line and the end point of the P wave.ECG recordings of at least 6 QRS for each lead 1 mV at a rate of 20 mm/s, including the complex 3 channels in amplitude and standard 12 leads will be done simultaneously.
P wave dispersion (PWD) | After the procedure of the fifteenth minute
  PWD in all leads will be measured manually with the X10 magnifying glass. The beginning of the P wave is the point where the isoelectric line and the P wave intersect. The endpoint was taken as the intersection of the isoelectric line and the end point of the P wave.ECG recordings of at least 6 QRS for each lead 1 mV at a rate of 20 mm/s, including the complex 3 channels in amplitude and standard 12 leads will be done simultaneously.
QTc (Corrected QT interval) and QTd (QT dispersion) values | Before the procedure
  The onset of the QRS complex and the descending T wave as the QT interval between the point where the arm cuts the isoelectric TP segment will be taken. QT dispersion (QTd) is the difference between the longest QT and the shortest QT interval. The heart rate-corrected value of the measurement of the QT interval will be used as the QTc. QTc > 500 ms means increased.
QTc (Corrected QT interval) and QTd (QT dispersion) values | After the procedure of the first minute
  The onset of the QRS complex and the descending T wave as the QT interval between the point where the arm cuts the isoelectric TP segment will be taken. QT dispersion (QTd) is the difference between the longest QT and the shortest QT interval. The heart rate-corrected value of the measurement of the QT interval will be used as the QTc. QTc > 500 ms means increased.
QTc (Corrected QT interval) and QTd (QT dispersion) values | After the procedure of the fifth minute
  The onset of the QRS complex and the descending T wave as the QT interval between the point where the arm cuts the isoelectric TP segment will be taken. QT dispersion (QTd) is the difference between the longest QT and the shortest QT interval. The heart rate-corrected value of the measurement of the QT interval will be used as the QTc. QTc > 500 ms means increased.
QTc (Corrected QT interval) and QTd (QT dispersion) values | After the procedure of the tenth minute
  The onset of the QRS complex and the descending T wave as the QT interval between the point where the arm cuts the isoelectric TP segment will be taken. QT dispersion (QTd) is the difference between the longest QT and the shortest QT interval. The heart rate-corrected value of the measurement of the QT interval will be used as the QTc. QTc > 500 ms means increased.
QTc (Corrected QT interval) and QTd (QT dispersion) values | After the procedure of the fifteenth minute
  The onset of the QRS complex and the descending T wave as the QT interval between the point where the arm cuts the isoelectric TP segment will be taken. QT dispersion (QTd) is the difference between the longest QT and the shortest QT interval. The heart rate-corrected value of the measurement of the QT interval will be used as the QTc. QTc > 500 ms means increased.

SECONDARY OUTCOMES:
Hospitalization | Before the procedure
  The diagnosis of all patients will be noted on the first day of the ICU.
Bronchoscopy duration | At the end of the procedure
  The duration of the procedure will be noted from the beginning of the bronchoscopy till the end of it.
Systolic blood pressure (SBP) | Before the procedure
  SBP will be measured from the monitor.
Systolic blood pressure (SBP) | After the procedure of the first minute
  SBP will be measured from the monitor.
Systolic blood pressure (SBP) | After the procedure of the fifth minute
  SBP will be measured from the monitor.
Systolic blood pressure (SBP) | After the procedure of the tenth minute
  SBP will be measured from the monitor.
Systolic blood pressure (SBP) | After the procedure of the fifteenth minute
  SBP will be measured from the monitor.
Diastolic blood pressure (DBP) | Before the procedure
  DBP will be measured from the monitor.
Diastolic blood pressure (DBP) | After the procedure of the first minute
  DBP will be measured from the monitor.
Diastolic blood pressure (DBP) | After the procedure of the fifth minute
  DBP will be measured from the monitor.
Diastolic blood pressure (DBP) | After the procedure of the tenth minute
  DBP will be measured from the monitor.
Diastolic blood pressure (DBP) | After the procedure of the fifteenth minute
  DBP will be measured from the monitor.
Mean arterial pressure (MAP) | Before the procedure
  The MAP is the average of the systolic pressure and the diastolic pressure that is formulized as MAP = (SBP + [2x DBP]) / 3.
Mean arterial pressure (MAP) | After the procedure of the first minute
  The MAP is the average of the systolic pressure and the diastolic pressure that is formulized as MAP = (SBP + [2x DBP]) / 3.
Mean arterial pressure (MAP) | After the procedure of the fifth minute
  The MAP is the average of the systolic pressure and the diastolic pressure that is formulized as MAP = (SBP + [2x DBP]) / 3.
Mean arterial pressure (MAP) | After the procedure of the tenth minute
  The MAP is the average of the systolic pressure and the diastolic pressure that formulized as MAP = (SBP + [2x DBP]) / 3.
Mean arterial pressure (MAP) | After the procedure of the fifteenth minute
  The MAP is the average of the systolic pressure and the diastolic pressure that is formulized as MAP = (SBP + [2x DBP]) / 3.
Heart rate (HR) | Before the procedure
  The HR value will be measured from the monitor.
Heart rate (HR) | After the procedure of the first minute
  The HR value will be measured from the monitor.
Heart rate (HR) | After the procedure of the fifth minute
  The HR value will be measured from the monitor.
Heart rate (HR) | After the procedure of the tenth minute
  The HR value will be measured from the monitor.
Heart rate (HR) | After the procedure of the fifteenth minute
  The HR value will be measured from the monitor.
Central venous pressure (CVP) | Before the procedure
  The CVP value will be measured from the monitor.
Central venous pressure (CVP) | After the procedure of the first minute
  The CVP value will be measured from the monitor.
Central venous pressure (CVP) | After the procedure of the fifth minute
  The CVP value will be measured from the monitor.
Central venous pressure (CVP) | After the procedure of the tenth minute
  The CVP value will be measured from the monitor.
Central venous pressure (CVP) | After the procedure of the fifteenth minute
  The CVP value will be measured from the monitor.
Peripheral oxygen saturation | Before the procedure
  This will be measured from the monitor.
Peripheral oxygen saturation | After the procedure of the first minute
  This will be measured from the monitor.
Peripheral oxygen saturation | After the procedure of the fifth minute
  This will be measured from the monitor.
Peripheral oxygen saturation | After the procedure of the tenth minute
  This will be measured from the monitor.
Peripheral oxygen saturation | After the procedure of the fifteenth minute
  This will be measured from the monitor.
Airway pressure (P Peak) | Before the procedure
  This will be measured from the monitor.
Airway pressure (P Peak) | After the procedure of the first minute
  This will be measured from the monitor.
Airway pressure (P Peak) | After the procedure of the fifth minute
  This will be measured from the monitor.
Airway pressure (P Peak) | After the procedure of the tenth minute
  This will be measured from the monitor.
Airway pressure (P Peak) | After the procedure of the fifteenth minute
  This will be measured from the monitor.
Respiratory rate | Before the procedure
  This will be measured from the monitor.
Respiratory rate | After the procedure of the first minute
  This will be measured from the monitor.
Respiratory rate | After the procedure of the fifth minute
  This will be measured from the monitor.
Respiratory rate | After the procedure of the tenth minute
  This will be measured from the monitor.
Respiratory rate | After the procedure of the fifteenth minute
  This will be measured from the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ozsari, Study Director — Abant İzzet Baysal Üniversitesi University
Locations (1):
- Abant izzet baysal university, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No